CLINICAL TRIAL: NCT02796859
Title: A Randomized Controlled Trial of Adjunctive Siltuximab in Schizophrenia
Brief Title: Siltuximab in Schizophrenia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brian Miller (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Brian Miller, Associate Professor, Augusta University
Organization: Augusta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15T-005
Record Dates: First submitted 2016-05-26; First posted 2016-06-13 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Inflammation; Psychosis; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Inflammation | interventions — siltuximab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Active Comparator): Subjects in the siltuximab group will receive an 11 mg/kg infusion at baseline, and weeks 3 and 6, as per the recommended dosing for multicentric Castleman's disease
  Interventions: Drug: Siltuximab
- Control Group (Placebo Comparator): Subjects in the placebo group will receive an infusion of normal saline (with the same packaging and volume as the siltuximab group) at baseline, and weeks 3 and 6.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Siltuximab — Investigational agent
  Other Names: Sylvant
  Arms: Treatment Group
Drug: normal saline — Placebo
  Other Names: 0.9% NS
  Arms: Control Group

SUMMARY:
This study is a Phase 1 clinical trial to determine the safety, tolerability, and efficacy of Siltuximab (Sylvant) as an adjunct to antipsychotic medications in stable outpatients with schizophrenia. Siltuximab (structural formula C6450H9932N1688O2016S50) is a recombinant chimeric (human-murine) anti-human interleukin-6 (IL-6) monoclonal antibody. Siltuximab is formulated as a concentrate for solution for infusion, and will be administered by intravenous infusion.

The investigators propose a 9-week randomized controlled trial of siltuximab, given in adjunct to antipsychotics, in N=30 stable outpatients with schizophrenia or schizoaffective disorder and evidence of increased inflammation in the peripheral blood (high-sensitivity C-reactive protein [hsCRP] >0.5 mg/dL). The investigators hypothesize that adjunctive treatment with siltuximab will be associated with significant improvement in cognition compared to placebo in patients with schizophrenia, baseline IL-6 levels are higher in siltuximab-treated responders versus non-responders, and there will be greater decreases in hsCRP from baseline to week 6 in siltuximab-treated versus placebo-treated responders, with response defined as ≥0.5 SD improvement in cognition. Siltuximab is administered as an intravenous infusion every 3 weeks. Following a screening evaluation, participants will receive three infusions of siltuximab, one at baseline, another at week 3 of the study, and another at week 6. The investigators will measure changes in cognitive function and symptoms over a 9-week period. Complementing previous positive clinical trials of non-steroidal anti-inflammatory drugs, this would be a "proof-of-concept" study that targeting specific cytokines is a viable treatment for schizophrenia.

Interleukin 6 and its receptor were discovered and cloned at Osaka University, Japan, by Tadamitsu Kishimoto in the 1980s. Janssen Pharmaceuticals, Inc. began the clinical development of siltuximab for the treatment of multicentric Castleman's disease, a rare blood disorder. Other clinical studies with siltuximab have been conduced for patients with B-cell non-Hodgkin's lymphoma, multiple myeloma, and ovarian cancer.

In April 2014,siltuxiumab was approved by the U.S. Food and Drug Administration (US FDA) as Sylvant for human immunodeficiency virus (HIV)-negative and human herpesvirus-8 (HHV-8)-negative multicentric Castleman's disease.

DETAILED DESCRIPTION:
A pathophysiological role for inflammation in schizophrenia has been one of the more enduring findings in the field. Recently, increased understanding of complex interactions between inflammation and the brain in other chronic diseases has better informed this relationship in schizophrenia. Several trials have found that treatment with non-steroidal anti-inflammatory drugs (NSAIDs), in adjunct to antipsychotics, was associated with significant improvement in psychopathology in schizophrenia. Cytokines are key regulators of inflammation that exert effects in the periphery and the brain. Serum cytokine levels predicted response in two studies , and another study found a trend for improved cognition with adjunctive NSAID treatment. These findings provide important empirical support for a pathophysiological role for inflammation in some patients with schizophrenia. Two important limitations of these trials are that: a) the agents investigated have relevant off-target (i.e., non-immune) effects, and b) evidence of inflammation in the peripheral blood was not an inclusion criterion, which may have decreased the signal-to-noise ratio.

Schizophrenia is associated with impaired cognition, which persists despite current treatments, and is an important determinant of quality of life and overall function. Converging lines of evidence suggest that interleukin-6 (IL-6) is a promising therapeutic target for cognitive impairment in schizophrenia. IL-6 is a cytokine produced by peripheral blood leukocytes, and central nervous system (CNS) microglia and astrocytes. The IL-6 gene is a risk factor for schizophrenia and may impact on serum IL-6 levels. Blood and cerebrospinal fluid (CSF) IL-6 levels are altered in schizophrenia. IL-6 levels are associated with psychopathology and cognition in schizophrenia. Serum IL-6 levels are also increased in prodromal psychosis, drug-naïve first-episode psychosis (FEP) and first-degree relatives of patients with schizophrenia. In populations outside of schizophrenia, higher serum IL-6 levels are associated with poorer cognition, cognitive decline, and smaller hippocampal volume. In FEP and chronic schizophrenia, IL-6 levels are a significant predictor of smaller left hippocampal volume.

Evidence from animal studies also supports a putative role for IL-6 in the pathophysiology of schizophrenia. A single maternal injection of IL-6 during mouse pregnancy caused prepulse and latent inhibition deficits in the adult offspring. In rat prenatal immune activation models, adult offspring have increased serum IL-6 levels, at an age with homology to the usual age of onset of schizophrenia, that are modulated by antipsychotics. Ketamine-induced neuronal production of IL-6 is responsible for the activation of brain N=nicotinamide adenine dinucleotide phosphate (NADPH)-oxidase and dysfunction of fast-spiking parvalbumin-expressing interneurons.

Along with our other previous work, our preliminary studies provide strong evidence that IL-6 is a novel therapeutic target for cognitive impairment in schizophrenia, and demonstrate the feasibility of the proposed trial. Briefly, in 64 patients with schizophrenia, the investigators found higher blood IL-6 levels were a significant predictor of greater impairment on the Brief Assessment of Cognition in Schizophrenia (BACS) after controlling for multiple potential confounding factors. In an 8-week open-label trial in 6 subjects, tocilizumab (an anti-IL-6 receptor monoclonal antibody), given in adjunct to antipsychotics, was well tolerated and associated with significant improvement in BACS verbal fluency at 4 weeks, BACS digit symbol coding at 2, 4, and 8 weeks, and BACS composite score at 4 and 8 weeks.

In the first year following the submission, one clinical trial is planned. The investigators will conduct a 9-week randomized, double-blind, placebo-controlled trial to determine the safety, tolerability, and efficacy of siltuximab as an adjunct to antipsychotic medications in 30 stable outpatients with schizophrenia.

Siltuximab has not been used before in the treatment of schizophrenia, and using it this way is experimental. The risks that have been found in people with multicentric Castleman's disease are known, but there may be unknown risks when used in schizophrenia. Clinically significant adverse drug reactions include anaphylaxis, renal failure, and pneumonia. Known side effects of siltuximab that are common include: swelling of the extremities, fatigue, itching, rash, weight gain, diarrhea, abdominal pain, and joint or limb pain. The most common side effect of the drug is nasopharyngitis, which occurs in 63% of subjects with long-term exposure to Siltuximab.

Subjects with schizophrenia and schizoaffective disorder will be accessed from outpatient psychiatry clinic at Augusta University or other satellite collaborative sites. The study has 5 visits: screening, baseline, and weeks 3, 6, and 9. Subjects will be randomized equally to either siltuximab (n=15) or placebo (n=15), in adjunct to their current antipsychotic and other psychotropic medications. The study has 5 visits: screening, baseline, and weeks 3, 6, and 9. Subjects will be randomized equally to either siltuximab (n=15) or placebo (n=15), in adjunct to their current antipsychotic and other psychotropic medications. Subjects in the siltuximab group will receive an 11 mg/kg infusion at baseline, and weeks 3 and 6, as per the recommended dosing for multicentric Castleman's disease. Subjects in the placebo group will receive an infusion of normal saline (with the same packaging and volume as the siltuximab group) at baseline, and weeks 3 and 6. Subjects will be monitored for an additional 30 minutes following the completion of the infusion. Dr. Miller will monitor the subject throughout the infusion and the 30 minute post-infusion period. The investigators will contact the subjects by phone on days 1 and 7 after each infusion to assess for any infusion-related events. The investigators will assess cognition and psychopathology at baseline, and at weeks 3, 6, and 9. The investigators will also measure a multiplex panel of blood cytokines (including IL-6) and tryptophan catabolites at baseline, and at weeks 3, 6, and 9. At Screening, all subjects will be administered the evaluation to sign consent, informed consent, and the structured clinical interview for Diagnostic and Statistical Manual of Mental Disorders (DSM) psychosis and affective disorders modules. The investigators will perform a medical history and physical exam, fasting labs (complete blood count [CBC], complete metabolic profile [CMP], hsCRP, lipid panel, urinalysis, and urine drug screen (UDS), hepatitis panel, HIV, rapid plasma reagin [RPR], and human chorionic gonadotropin [hCG] in females), a tuberculin skin test, and a 12-lead electrocardiogram. At Baseline, the investigators will perform the Positive And Negative Syndrome Scale (PANSS), BACS, and Clinical Global Impressions scale (CGI), Calgary Depression Scale (CDS) and Short Form Health Survey (SF-36) and draw blood for IL-6 and high-sensitivity c-reactive protein (hsCRP). At Week 3, 6, and 9, the investigators will perform an interval history, physical exam, PANSS, BACS, CGI, CDS, SF-36, and obtain fasting labs (CBC, CMP, lipid panel, hsCRP, urinalysis, UDS, and hCG in females). Different versions of the BACS will be used to avoid practice effects. Patients will be withdrawn if they meet any exclusion criterion at any time point.

ELIGIBILITY:
Inclusion Criteria:

* capable of giving informed consent
* diagnosis of schizophrenia or schizoaffective disorder
* stable based on clinical judgment
* taking a non-clozapine antipsychotic
* on the same psychotropic medications for >4 weeks
* hsCRP >0.3 mg/dL at the screening visit

Exclusion Criteria:

* imminent danger to self/others
* antibiotic use in the past 2 weeks
* current scheduled use of immunomodulatory agents
* history of an immune disorder
* illicit drug use in the past 30 days
* any unstable or untreated medical condition
* history of gastrointestinal ulcers, diverticulitis, malignancy, CNS demyelinating disorder, seizure disorder, or exposure to tuberculosis
* low absolute neutrophil (<2000) or platelet (<100,000) count
* abnormal hepatic function (AST or ALT >1.5 times the upper limit of normal) or renal function (BUN or creatinine >1.5 times the upper limit of normal)
* any abnormal lab test result judged to be clinically significant
* active or chronic infections
* pregnancy, breast feeding, or female of child-bearing potential who is not using any contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition | Baseline and 9 weeks
  The Brief Assessment of Cognition in Schizophrenia (BACS) is the metric used to characterize cognition in this study. The BACS consists of 6 subscales: Verbal Memory (range 0-75), Working Memory (range 0-28), Motor Speed (range 0-100), Verbal Fluency (measure is total number of words generated in two 60 second trials), Attention and Processing speed (range 0-110), and Executive Function (range 0-22). For each subscale, higher scores reflect better cognition. For each subscale, a Standard Deviation Score was calculated based on normative data (Keefe et al. Norms and standardization of the Brief Assessment of Cognition in Schizophrenia (BACS). Schizophrenia Research 102 (2008) 108-115). The BACS composite score is calculated as the average Standard Deviation Score of the 6 subscale scores. The change in BACS composite score will be calculated as the BACS composite score at 9 weeks minus the BACS composite score at baseline.

SECONDARY OUTCOMES:
Change in Total Psychotic Symptoms | Baseline and 9 weeks
  The Positive and Negative Symptoms Scale (PANSS) is the metric used to characterize psychotic symptoms in this study. The PANSS consists of 30 items, each scored 1-7. The range for the PANSS total score is 30-210. There are 3 subscales - PANSS positive score (range 7-49), PANSS negative score (range 7-49), and PANSS general score (range 16-112). PANSS total score is the summation of these 3 subscales. Higher values for the total and subscale scores reflect more severe psychopathology. A positive change in PANSS total score reflects an increase in psychopathology. A negative change in PANSS total score reflects a decrease in psychopathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Muller N. COX-2 inhibitors as antidepressants and antipsychotics: clinical evidence. Curr Opin Investig Drugs. 2010 Jan;11(1):31-42. PMID 20047157
- [Background] Muller N, Krause D, Dehning S, Musil R, Schennach-Wolff R, Obermeier M, Moller HJ, Klauss V, Schwarz MJ, Riedel M. Celecoxib treatment in an early stage of schizophrenia: results of a randomized, double-blind, placebo-controlled trial of celecoxib augmentation of amisulpride treatment. Schizophr Res. 2010 Aug;121(1-3):118-24. doi: 10.1016/j.schres.2010.04.015. Epub 2010 May 31. PMID 20570110
- [Background] Nitta M, Kishimoto T, Muller N, Weiser M, Davidson M, Kane JM, Correll CU. Adjunctive use of nonsteroidal anti-inflammatory drugs for schizophrenia: a meta-analytic investigation of randomized controlled trials. Schizophr Bull. 2013 Nov;39(6):1230-41. doi: 10.1093/schbul/sbt070. Epub 2013 May 29. PMID 23720576
- [Background] Sommer IE, van Westrhenen R, Begemann MJ, de Witte LD, Leucht S, Kahn RS. Efficacy of anti-inflammatory agents to improve symptoms in patients with schizophrenia: an update. Schizophr Bull. 2014 Jan;40(1):181-91. doi: 10.1093/schbul/sbt139. Epub 2013 Oct 8. PMID 24106335
- [Background] Muller N, Ulmschneider M, Scheppach C, Schwarz MJ, Ackenheil M, Moller HJ, Gruber R, Riedel M. COX-2 inhibition as a treatment approach in schizophrenia: immunological considerations and clinical effects of celecoxib add-on therapy. Eur Arch Psychiatry Clin Neurosci. 2004 Feb;254(1):14-22. doi: 10.1007/s00406-004-0478-1. PMID 14991374
- [Background] Laan W, Grobbee DE, Selten JP, Heijnen CJ, Kahn RS, Burger H. Adjuvant aspirin therapy reduces symptoms of schizophrenia spectrum disorders: results from a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2010 May;71(5):520-7. doi: 10.4088/JCP.09m05117yel. PMID 20492850
- [Background] Muller N, Riedel M, Schwarz MJ, Engel RR. Clinical effects of COX-2 inhibitors on cognition in schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2005 Apr;255(2):149-51. doi: 10.1007/s00406-004-0548-4. Epub 2004 Nov 19. PMID 15549344
- [Background] Paul-Samojedny M, Kowalczyk M, Suchanek R, Owczarek A, Fila-Danilow A, Szczygiel A, Kowalski J. Functional polymorphism in the interleukin-6 and interleukin-10 genes in patients with paranoid schizophrenia--a case-control study. J Mol Neurosci. 2010 Sep;42(1):112-9. doi: 10.1007/s12031-010-9365-6. PMID 20393813
- [Background] Sun S, Wang F, Wei J, Cao LY, Qi LY, Xiu MH, Chen S, Li XH, Kosten TA, Kosten TR, Zhang XY. Association between interleukin-6 receptor polymorphism and patients with schizophrenia. Schizophr Res. 2008 Jul;102(1-3):346-7. doi: 10.1016/j.schres.2008.04.018. Epub 2008 May 27. No abstract available. PMID 18508242
- [Background] Miller BJ, Buckley P, Seabolt W, Mellor A, Kirkpatrick B. Meta-analysis of cytokine alterations in schizophrenia: clinical status and antipsychotic effects. Biol Psychiatry. 2011 Oct 1;70(7):663-71. doi: 10.1016/j.biopsych.2011.04.013. Epub 2011 Jun 8. PMID 21641581
- [Background] Garver DL, Tamas RL, Holcomb JA. Elevated interleukin-6 in the cerebrospinal fluid of a previously delineated schizophrenia subtype. Neuropsychopharmacology. 2003 Aug;28(8):1515-20. doi: 10.1038/sj.npp.1300217. Epub 2003 Jun 11. PMID 12799618
- [Background] Sasayama D, Hattori K, Wakabayashi C, Teraishi T, Hori H, Ota M, Yoshida S, Arima K, Higuchi T, Amano N, Kunugi H. Increased cerebrospinal fluid interleukin-6 levels in patients with schizophrenia and those with major depressive disorder. J Psychiatr Res. 2013 Mar;47(3):401-6. doi: 10.1016/j.jpsychires.2012.12.001. Epub 2013 Jan 3. PMID 23290488
- [Background] Krause DL, Wagner JK, Wildenauer A, Matz J, Weidinger E, Riedel M, Obermeier M, Gruber R, Schwarz M, Muller N. Intracellular monocytic cytokine levels in schizophrenia show an alteration of IL-6. Eur Arch Psychiatry Clin Neurosci. 2012 Aug;262(5):393-401. doi: 10.1007/s00406-012-0290-2. Epub 2012 Jan 21. PMID 22271344
- [Background] Frydecka D, Misiak B, Pawlak-Adamska E, Karabon L, Tomkiewicz A, Sedlaczek P, Kiejna A, Beszlej JA. Interleukin-6: the missing element of the neurocognitive deterioration in schizophrenia? The focus on genetic underpinnings, cognitive impairment and clinical manifestation. Eur Arch Psychiatry Clin Neurosci. 2015 Sep;265(6):449-59. doi: 10.1007/s00406-014-0533-5. Epub 2014 Sep 12. PMID 25214388
- [Background] Miller B, Mellor A, Buckley PF. Interleukin-6 and Cognition in Non-Affective Psychosis. Schizophrenia Bulletin 2013(39): S242-S243.
- [Background] Stojanovic A, Martorell L, Montalvo I, Ortega L, Monseny R, Vilella E, Labad J. Increased serum interleukin-6 levels in early stages of psychosis: associations with at-risk mental states and the severity of psychotic symptoms. Psychoneuroendocrinology. 2014 Mar;41:23-32. doi: 10.1016/j.psyneuen.2013.12.005. Epub 2013 Dec 14. PMID 24495605
- [Background] Nunes SO, Matsuo T, Kaminami MS, Watanabe MA, Reiche EM, Itano EN. An autoimmune or an inflammatory process in patients with schizophrenia, schizoaffective disorder, and in their biological relatives. Schizophr Res. 2006 May;84(1):180-2. doi: 10.1016/j.schres.2006.02.003. Epub 2006 Mar 10. No abstract available. PMID 16530388
- [Background] Elderkin-Thompson V, Irwin MR, Hellemann G, Kumar A. Interleukin-6 and memory functions of encoding and recall in healthy and depressed elderly adults. Am J Geriatr Psychiatry. 2012 Sep;20(9):753-63. doi: 10.1097/JGP.0b013e31825d08d6. PMID 22892560
- [Background] Sasayama D, Hori H, Teraishi T, Hattori K, Ota M, Matsuo J, Kawamoto Y, Kinoshita Y, Amano N, Kunugi H. Association of cognitive performance with interleukin-6 receptor Asp358Ala polymorphism in healthy adults. J Neural Transm (Vienna). 2012 Mar;119(3):313-8. doi: 10.1007/s00702-011-0709-3. Epub 2011 Aug 31. PMID 21879314
- [Background] Frodl T, Carballedo A, Hughes MM, Saleh K, Fagan A, Skokauskas N, McLoughlin DM, Meaney J, O'Keane V, Connor TJ. Reduced expression of glucocorticoid-inducible genes GILZ and SGK-1: high IL-6 levels are associated with reduced hippocampal volumes in major depressive disorder. Transl Psychiatry. 2012 Mar 13;2(3):e88. doi: 10.1038/tp.2012.14. PMID 22832853
- [Background] Marsland AL, Petersen KL, Sathanoori R, Muldoon MF, Neumann SA, Ryan C, Flory JD, Manuck SB. Interleukin-6 covaries inversely with cognitive performance among middle-aged community volunteers. Psychosom Med. 2006 Nov-Dec;68(6):895-903. doi: 10.1097/01.psy.0000238451.22174.92. PMID 17132839
- [Background] Marsland AL, Gianaros PJ, Abramowitch SM, Manuck SB, Hariri AR. Interleukin-6 covaries inversely with hippocampal grey matter volume in middle-aged adults. Biol Psychiatry. 2008 Sep 15;64(6):484-90. doi: 10.1016/j.biopsych.2008.04.016. Epub 2008 Jun 2. PMID 18514163
- [Background] Kalmady SV, Venkatasubramanian G, Shivakumar V, Gautham S, Subramaniam A, Jose DA, Maitra A, Ravi V, Gangadhar BN. Relationship between Interleukin-6 gene polymorphism and hippocampal volume in antipsychotic-naive schizophrenia: evidence for differential susceptibility? PLoS One. 2014 May 2;9(5):e96021. doi: 10.1371/journal.pone.0096021. eCollection 2014. PMID 24787542
- [Background] Miller BJ, Timonen M, Isohanni M. Cytokine abnormalities, inflammation and psychosis in the northern Finland 1966 birth cohort. European Psychiatry 2014 (29): S519.
- [Background] Mondelli V, Cattaneo A, Murri MB, Di Forti M, Handley R, Hepgul N, Miorelli A, Navari S, Papadopoulos AS, Aitchison KJ, Morgan C, Murray RM, Dazzan P, Pariante CM. Stress and inflammation reduce brain-derived neurotrophic factor expression in first-episode psychosis: a pathway to smaller hippocampal volume. J Clin Psychiatry. 2011 Dec;72(12):1677-1684. doi: 10.4088/JCP.10m06745. Epub 2011 May 18. PMID 21672499
- [Background] Smith SE, Li J, Garbett K, Mirnics K, Patterson PH. Maternal immune activation alters fetal brain development through interleukin-6. J Neurosci. 2007 Oct 3;27(40):10695-702. doi: 10.1523/JNEUROSCI.2178-07.2007. PMID 17913903
- [Background] Basta-Kaim A, Szczesny E, Leskiewicz M, Glombik K, Slusarczyk J, Budziszewska B, Regulska M, Kubera M, Nowak W, Wedzony K, Lason W. Maternal immune activation leads to age-related behavioral and immunological changes in male rat offspring - the effect of antipsychotic drugs. Pharmacol Rep. 2012;64(6):1400-10. doi: 10.1016/s1734-1140(12)70937-4. PMID 23406750
- [Background] Romero E, Ali C, Molina-Holgado E, Castellano B, Guaza C, Borrell J. Neurobehavioral and immunological consequences of prenatal immune activation in rats. Influence of antipsychotics. Neuropsychopharmacology. 2007 Aug;32(8):1791-804. doi: 10.1038/sj.npp.1301292. Epub 2006 Dec 20. PMID 17180123
- [Background] Romero E, Guaza C, Castellano B, Borrell J. Ontogeny of sensorimotor gating and immune impairment induced by prenatal immune challenge in rats: implications for the etiopathology of schizophrenia. Mol Psychiatry. 2010 Apr;15(4):372-83. doi: 10.1038/mp.2008.44. Epub 2008 Apr 15. PMID 18414405
- [Background] Behrens MM, Ali SS, Dugan LL. Interleukin-6 mediates the increase in NADPH-oxidase in the ketamine model of schizophrenia. J Neurosci. 2008 Dec 17;28(51):13957-66. doi: 10.1523/JNEUROSCI.4457-08.2008. PMID 19091984
- [Background] Miller BJ, Culpepper N, Rapaport MH. C-reactive protein levels in schizophrenia: a review and meta-analysis. Clin Schizophr Relat Psychoses. 2014 Jan;7(4):223-30. PMID 23428789
- [Background] Miller BJ, Mellor A, Buckley P. Total and differential white blood cell counts, high-sensitivity C-reactive protein, and the metabolic syndrome in non-affective psychoses. Brain Behav Immun. 2013 Jul;31:82-9. doi: 10.1016/j.bbi.2012.08.016. Epub 2012 Sep 11. PMID 22982547
- [Background] Miller BJ, Kandhal P, Rapaport MH, Mellor A, Buckley P. Total and differential white blood cell counts, high-sensitivity C-reactive protein, and cardiovascular risk in non-affective psychoses. Brain Behav Immun. 2015 Mar;45:28-35. doi: 10.1016/j.bbi.2014.12.005. Epub 2014 Dec 24. PMID 25542737
- [Background] Miller BJ, Dias JK, Lemos HP, Buckley PF. An open-label, pilot trial of adjunctive tocilizumab in schizophrenia. J Clin Psychiatry. 2016 Feb;77(2):275-6. doi: 10.4088/JCP.15l09920. No abstract available. PMID 26930525